CLINICAL TRIAL: NCT04476810
Title: Long Term Outcome of Combined Phacoemulsification and Excisional Goniotomy With the Kahook Dual Blade
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Al Habash (Other)
Responsible Party: Sponsor-Investigator, Ahmed Al Habash, Dr. Ahmed Al Habash, MD assistant professor, consultant cataract and glaucoma, Imam Abdulrahman Bin Faisal University
Organization: Imam Abdulrahman Bin Faisal University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB -2020-01-169
Record Dates: First submitted 2020-07-10; First posted 2020-07-20 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Glaucoma; Glaucoma, Open-Angle; Cataract; Angle Closure Glaucoma; Surgery
Keywords: glaucoma; goniotomy; Kahook Dual Blade; combined phacoemulsification; MIGS; Schlemm's Canal
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle; Cataract; Glaucoma, Angle-Closure | interventions — Phacoemulsification

STUDY DESIGN:
Intervention Model Description: Prospective, non-comparative, uncontrolled, non-randomized interventional case series. Consecutive patients with medically-treated glaucoma and visually-significant cataract underwent combined surgery. Subgroup analysis of glaucoma subtypes was performed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- combined (phaco-kdb) (Experimental): Prospective, non-comparative, uncontrolled, non-randomized interventional case series. Consecutive patients with medically-treated glaucoma and visually-significant cataract underwent combined surgery. Subgroup analysis of glaucoma subtypes was performed.
  Interventions: Device: kahook dual blade

INTERVENTIONS:
Device: kahook dual blade — Combined Phacoemulsification and Excisional Goniotomy with the Kahook Dual Blade
  Other Names: phacoemulsification

SUMMARY:
Purpose: Characterize changes in intraocular pressure (IOP), IOP-lowering medications, and visual acuity (VA) through 3 years in patients undergoing combined phacoemulsification and excisional goniotomy with the Kahook Dual Blade (phaco-KDB), with simultaneous goniosynechialysis in cases of angle-closure glaucoma, by a single surgeon (A.H.) in King Fahd Hospital of the University, Dammam, Saudi Arabia.

Methods: Prospective, non-comparative, uncontrolled, non-randomized interventional case series. Consecutive patients with medically-treated glaucoma and visually-significant cataract underwent combined surgery. Subgroup analysis of glaucoma subtypes was performed.

ELIGIBILITY:
inclusion criteria:

* adults 18 years or older
* medically-managed glaucoma
* visually significant cataract

Exclusion Criteria:

* Patients undergoing any other combined procedures
* active uveitis
* coexisting retinopathy that limits visual acuity potential
* active neovascularization
* angle dysgenesis
* those with less than 6 months of follow-up, were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure | 36 months
  Characterize changes in intraocular pressure (IOP) in mmHg goldmann applanation tonometry each visit in the clinic after the combined phacoemulsification and excisional goniotomy with the kahook dual blade.
Intraocular pressure lowering medications | 36 months
  count the change in number of Intraocular pressure lowering medications each visit in the clinic after the combined phacoemulsification and excisional goniotomy with the kahook dual blade

SECONDARY OUTCOMES:
Visual acuity | 36 months
  Characterize visual acuity (VA) using logMAR chart, each visit in clinic post undergoing combined phacoemulsification and excisional goniotomy with the kahook dual blade.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Al habash, MD, Principal Investigator — assistant professor
Locations (1):
- Imam Abdulrahman Bin Faisal University Hospital, Dammam, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided